CLINICAL TRIAL: NCT03041688
Title: A Phase 1B Study of KRT-232 (AMG-232) in Combination With Decitabine and Venetoclax in Acute Myeloid Leukemia
Brief Title: Testing a New Chemotherapy Drug, KRT-232 (AMG-232) in Combination With Decitabine and Venetoclax in Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-00128; NCI-2017-00128 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-92; 10075 (Other: City of Hope Comprehensive Cancer Center LAO); 10075 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Decitabine; Injections; navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; 2-(5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-(1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, navtemadlin, venetoclax) (Experimental): Patients receive decitabine IV over 1 hour on days 1-10, navtemadlin PO QD on days 1-7, and venetoclax PO QD on days 1-21. Treatment repeats every 28 days for up to 4 cycles in patients with evidence of persistent AML.
  Starting cycle 2, patients with no morphologic evidence of AML receive decitabine IV over 1 hour on days 1-5, navtemadlin PO QD on days 1-7, and venetoclax PO QD on days 1-14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients also undergo bone marrow aspiration and biopsy, and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine; Drug: Navtemadlin; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Navtemadlin — Given PO
  Other Names: (3R,5R,6S)-5-(3-Chlorophenyl)-6-(4-chlorophenyl)-3-methyl-1-((1S)-2-methyl-1-(((1-methylethyl)sulfonyl)methyl)propyl)-2-oxo-3-piperidineacetic Acid; AMG 232; AMG-232; KRT 232; KRT-232; KRT232; MDM2 Inhibitor KRT-232
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase Ib trial studies the side effects and best dose of navtemadlin when given together with decitabine and venetoclax in treating patients with acute myeloid leukemia that has come back after a period of improvement (recurrent), does not respond to treatment (refractory), or is newly diagnosed. Navtemadlin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving navtemadlin, decitabine, and venetoclax together may work better than decitabine alone in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the toxicities of navtemadlin (KRT-232 [AMG-232]) in combination with decitabine (20 mg/m^2 for 10 days), and venetoclax, and to determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of KRT-232 (AMG-232) in combination with a standard dose of decitabine and venetoclax.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetic (PK) profiles of KRT-232 (AMG-232), venetoclax, and decitabine when used in combination.

II. To evaluate p53 signaling induced by KRT-232 (AMG-232), venetoclax, and decitabine as measured by MIC-1 induction.

III. To correlate KRT-232 (AMG-232), venetoclax and decitabine exposure with pharmacodynamics endpoints (efficacy, toxicity, changes in p53 signaling).

EXPLORATORY OBJECTIVES:

I. To evaluate the response rate (RR) and progression free survival (PFS) of KRT-232 (AMG-232), venetoclax, and decitabine in acute myeloid leukemia (AML).

II. To evaluate potential predictive biomarkers of response to KRT-232 (AMG-232), venetoclax, and decitabine in AML.

III. To evaluate the pharmacodynamic (PD) effects of KRT-232 (AMG-232), venetoclax and decitabine in AML blasts.

IV. To determine the variability of decitabine incorporation into genomic deoxyribonucleic acid (DNA) and correlate with systemic pharmacokinetics and exposure-response relationships.

OUTLINE: This is a dose-escalation study of navtemadlin.

Patients receive decitabine intravenously (IV) over 1 hour on days 1-10, navtemadlin orally (PO) once daily (QD) on days 1-7, and venetoclax PO QD on days 1-21. Treatment repeats every 28 days for up to 4 cycles in patients with evidence of persistent AML.

Starting cycle 2, patients with no morphologic evidence of AML receive decitabine IV over 1 hour on days 1-5, navtemadlin PO QD on days 1-7, and venetoclax PO QD on days 1-14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients also undergo bone marrow aspiration and biopsy, and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory AML (>= 5% blasts in bone marrow or extramedullary leukemia); adverse cytogenetics, e.g., as defined by the Medical Research Council (MRC) Prognostic Groupings; secondary AML; organ dysfunction arising from significant co-morbidities not directly linked to leukemia; Eastern Cooperative Oncology Group [ECOG] = 2) or not willing to undergo intensive chemotherapy
* Patients must have measurable disease as defined the presence of >= 20% blasts in bone marrow or extramedullary leukemia
* Eligible patient must show evidence of wild-type (WT) p53 as assessed by DNA sequencing; note, that since patients with AML have a rapidly proliferating disease, patient can be enrolled and begin treatment prior to obtaining the results of this test; patients who are found to the TP53 mutated will be removed from study and can continue on single agent decitabine; however patients will continue to be followed for toxicity
* Age >= 18 years; because no dosing or adverse event data are currently available on the use of KRT-232 (AMG-232) in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* ECOG performance status =< 2 (Karnofsky >= 60%)
* White blood count =< 25 x 10^9/L
* Total bilirubin < 1.5 x institutional upper limit of normal (ULN) (< 2.0 x ULN for subjects with documented Gilbert's syndrome or < 3.0 x ULN for subjects for whom the indirect bilirubin level suggests an extrahepatic source of elevation)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN
* Alkaline phosphatase < 2.0 x ULN (if liver or bone metastases are present, < 3.0 x ULN)
* Body surface area (BSA)-normalized creatinine clearance >= 30 mL/min/1.73 m^2 (using Cockcroft-Gault creatinine clearance [CrCl])
* Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN), OR international normalized ratio (INR) < 1.5
* Patient must be willing to submit the blood sampling and bone marrow sampling for the PK and PD analyses and exploratory biomarkers
* The effects of KRT-232 (AMG-232) on the developing human fetus are unknown; for this reason and because decitabine is known to be teratogenic, women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation through 5 weeks (women) after receiving the last dose of KRT-232 (AMG-232); should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of KRT-232 (AMG-232) administration

  * Adequate methods of effective birth control include sexual abstinence (men, women); vasectomy; or a condom with spermicide (men) in combination with barrier methods, hormonal birth control or intrauterine device (IUD) (women)
* Ability to understand and the willingness to sign a written informed consent document
* White blood cell (WBC) count =< 25,000/uL before administration of decitabine on cycle 1 day 1; Note: hydroxyurea may be used to control the level of circulating leukemic blast cell counts to not lower than 10,000/uL during the study

Exclusion Criteria:

* Acute promyelocytic leukemia with t(15;17)(q22;q12) and/or PML-RARA molecular rearrangement
* Patients with previously untreated AML with core binding factor (CBF) chromosomal aberrations (inv[16]/t[16;16] or t[8;21]); Note that patients with relapsed or refractory AML with CBF chromosomal aberrations will be eligible
* Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 0 or 1, or to levels dictated in the eligibility criteria with the exception of alopecia (grade 2 or 3 toxicities from prior antitumor therapy that are considered irreversible [defined as having been present and stable for > 6 months], such as ifosfamide-related proteinuria, may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and sponsor)
* Patients who are receiving any other investigational agents
* Major surgery within 28 days of study day 1
* Patients with known central nervous system involvement at the time of study entry will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to KRT-232 (AMG-232) or decitabine
* All herbal medicines (e.g., St. John's wort), vitamins, and supplements consumed by the subject within the 30 days prior to receiving the first dose of KRT-232 (AMG-232) or venetoclax, and continuing use, if applicable, will be reviewed by the principal investigator
* Avoid and seek alternatives to the use of KRT-232 with sensitive substrates of CYP3A. If use of a sensitive CYP3A substrate with KRT-232 cannot be avoided, monitor subjects closely for toxicity. There is no identified drug-drug interaction potential for KRT-232 with other CYP enzymes
* Patient must not have received known moderate or strong CYP3A inducers within 7 days of enrollment; antifungal drugs, including those that are CYP3A inhibitors, are permitted; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Treatment with medications known to cause corrected QT (QTc) interval prolongation within 7 days of study day 1 is not permitted unless approved by the principal investigator; use of ondansetron is permitted for treatment of nausea and vomiting
* Current use of warfarin, factor Xa inhibitors and direct thrombin inhibitors

  * Note: Low molecular weight heparin and prophylactic low dose warfarin are permitted; PT/PTT must meet the inclusion criteria; subjects taking warfarin must have their INR followed closely
* Uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients receiving an anti-microbial agent may be eligible if the patient remains afebrile and hemodynamically stable for 72 hours; patients with myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association [NYHA] class III and higher), unstable angina, or cardiac arrhythmia requiring medication are excluded
* Patients with gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
* Patients with history of bleeding diathesis
* Positive hepatitis B surface antigen (HepBsAg) (indicative of chronic hepatitis B), positive hepatitis total core antibody with negative HBsAG (suggestive of occult hepatitis B), or detectable hepatitis C virus ribonucleic acid (RNA) by a polymerase-chain reaction (PCR) assay (indicative of active hepatitis C - screening is generally done by hepatitis C antibody [HepCAb], followed by hepatitis C virus RNA by PCR if HepCAb is positive)
* Human immunodeficiency virus (HIV)-patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based test
* Men and women of reproductive potential who are unwilling to practice acceptable methods of effective birth control while on study through 5 weeks (women) or 3 months and 1 week (men) after receiving the last dose of KRT-232 (AMG-232); acceptable methods of effective birth control include sexual abstinence (men, women); vasectomy; or a condom with spermicide (men) in combination with barrier methods, hormonal birth control or IUD (women)
* Pregnant women are excluded from this study because KRT-232 (AMG-232) is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with KRT-232 (AMG-232), breastfeeding should be discontinued if the mother is treated with KRT-232 (AMG-232); these potential risks may also apply to other agents used in this study
* Patients with a baseline QTc > 500 msec and patients with a family history of prolonged QT syndrome
* Patients with known TP53 mutations or chromosome 17 or 17p deletions
* Patients previously treated with azacytidine, decitabine, or venetoclax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-02-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity | Up to 4 weeks
  Will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) will be determined. Based on the toxicity observed, a derived variable, the occurrence of dose limiting toxicity, will be created. Will be correlated with MDM2 Inhibitor KRT-232 (KRT-232) (MDM2 inhibitor AMG-232 [AMG-232]) and decitabine exposure. Toxicities will be tabulated and reported according to dose level, grade, type, cycle, and attribution- and, if numbers permit, by whether the patient had newly diagnosed or previously treated acute myeloid leukemia (AML). Cumulative incidence curves will be used to estimate the proportion of patients who will discontinue therapy for reasons of toxicity or general inability to tolerate the regimen. The data from all patients treated at the RP2D, will be combined for a final summary and listing of toxicities observed.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) profile | Baseline, 1, 3, 5, 8 and 24 hours post dose on days 4 and 18 of course 1; baseline, 0.5 hour, prior to end of infusion, 0.25, 0.5, and 1 hour post infusion on days 1 and 4 of course 1
  Will be measured using liquid chromatography/tandem mass spectrometric method. Standard descriptive methods (point estimates and confidence intervals, scatterplots) will be used to summarize the baseline levels and the changes from baseline (i.e. after treatment). The individual PK parameters from a single dose will be estimated maximum concentration (Cmax), area under the curve (AUC), half-life (T1/2), apparent clearance, and apparent volume of distribution using non-compartmental or compartmental PK methods with the software WinNonlin. Cmax and AUC will be calculated for decitabine systemic exposure.
P53 activation | Up to 4 weeks
  Will be measured by MIC-1 levels. For serum MIC-1 levels, each individual level will be normalized to the baseline level for that patient. Will be analyzed using nonparametric statistics. Significance for comparisons will be at the p < 0.05 level.
Change in p53 signaling | Baseline to 30 days after end of study treatment
  Will be correlated with KRT-232 (AMG-232) and decitabine exposure. Will be analyzed using nonparametric statistics. Significance for comparisons will be at the p < 0.05 level.

OTHER OUTCOMES:
Complete response (CR) or CR with incomplete blood count recovery | Up to 112 days
  The percent of CR's will be calculated and associated exact 95% confidence intervals will be constructed.
Complete cytogenetic response (CRc or molecular CR [CRm]) | Up to 112 days
  Will be evaluated according to revised International Working Group criteria. The percent of CR's will be calculated and associated exact 95% confidence intervals will be constructed.
Progression-free survival (PFS) | From start of treatment to progression/recurrence or death, whichever comes first, assessed up to 4 weeks
  Kaplan-Meier plots will be used to summarize PFS.
Pharmacodynamic (PD) effects on leukemia blasts | Up to 4 weeks
  PD effects of KRT-232 (AMG-232) in combination with decitabine on leukemia blasts will be explored.
Predictive biomarker of sensitivity | Up to 4 weeks
  PD effects of KRT-232 (AMG-232) in combination with decitabine on potential predictive biomarker of sensitivity will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Kelly, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (13):
- United States (13):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia